CLINICAL TRIAL: NCT01187524
Title: The Natural History of Reproductive and Overall Health in Women With a Pre-Mutation in the FMR1 Gene: Creation of a Patient Registry
Brief Title: The Natural History of Reproductive and Overall Health in Girls and Women With a Pre-Mutation in the FMR1 Gene; Creation of a Patient Registry
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100144; 10-CH-0144
Record Dates: First submitted 2010-08-21; First posted 2010-08-24 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-05-31

CONDITIONS: Fragile X Syndrome; FMR1 Premutation; Primary Ovairan Insufficiency; Premature Ovarian Failure; Premature Menopause
Keywords: Patient Registry; FMR1 Gene; Fragile X Syndrome; Primary Ovarian Insufficiency; Premature Ovarian Failure; Premature Ovarian Insufficiency
MeSH Terms: conditions — Fragile X Syndrome; Primary Ovarian Insufficiency; Menopause, Premature

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* In human DNA, the Fragile X (FMR1) gene helps to regulate the nervous and reproductive systems. If the gene is abnormal, it can cause different kinds of problems, such as abnormal menstrual periods, decreased fertility, muscle tremors, and mental retardation. An abnormal FMR1 gene can also make a person more susceptible to other medical conditions, such as thyroid problems, high blood pressure, seizures, and depression. More research is needed on how abnormalities in the FMR1 gene can lead to these problems, and how often these problems appear in individuals with an abnormal FMR1 gene.
* Researchers are interested in developing a patient registry of women who have an abnormality in the FMR1 gene. This registry will allow researchers to follow participants over time and study possible effects of this abnormality on their general and reproductive health.

Objectives:

- To develop a patient registry of women with an abnormal FMR1 gene and monitor their general and reproductive health.

Eligibility:

- Women at least 18 years of age who have an abnormal FMR1 gene on the X chromosome.

Design:

* The following groups of women will be eligible for screening for this study:
* Those who have a family member with Fragile X Syndrome or mental retardation
* Those who have (or have a family member who has) primary ovarian insufficiency, also known as premature menopause
* Those who have (or have a family member who has) certain neurological problems such as tremors or Parkinson's disease.
* Eligible participants will be scheduled for an initial study visit at the National Institutes of Health Clinical Center. Participants who have regular menstrual periods should schedule the visit between days 3 and 8 of the menstrual cycle; those who do not have regular periods may have the visit at any time of the month. In addition, all estrogen-based treatments (such as birth control pills) must be stopped for 2 weeks prior to the study visit.
* Participants will have a full physical examination, provide a medical history, and provide blood samples for immediate and future testing. Participants will return for yearly visits for the same tests for as long as the study continues.
* Participants who have or develop primary ovarian insufficiency related to the FMR1 gene will also have tests to measure bone thickness and will have a vaginal ultrasound to examine the ovaries. These tests will be scheduled for a separate visit, and will be repeated every 5 years for the duration of the study.

DETAILED DESCRIPTION:
Spontaneous 46,XX primary ovarian insufficiency (POI) is a cause of decreased fertility in approximately 1% of women before age 40. The most common known genetic cause of 46,XX POI is a pre -mutation in the Fragile X Mental Retardation (FMR1) gene. The FMR1 gene is located on the X-chromosome and contains a CGG repeat in the un-translated region; this CGG repeat is normally present in less than 55 copies, but has a tendency to expand across generations. Greater than 200 CGG copies results in Fragile X Syndrome (FXS), the most common form of heritable mental retardation. A pre-mutation in the FMR1 gene, defined as between 55 and 199 CGG repeats, is associated with POI in women and carries a risk of expanding to the full mutation in a woman s offspring, resulting in a child with FXS. POI that is associated with the FMR1 pre-mutation is known as Fragile X-associated POI ( FXPOI ). Approximately 20% of women with an FMR1 pre-mutation develop FXPOI. Importantly, it is not known why some women with the pre-mutation develop FXPOI and others do not. The primary objective of this study is to characterize the natural history of reproductive function in women who are FMR1 pre-mutation carriers by creating a patient registry that will allow us to follow them longitudinally. Given the relative rarity of this pre-mutation in the general population (<1%), a patient registry is necessary for enrollment of an adequate number of patients for clinically significant analyses to be performed.

In order to characterize the natural history of reproductive function in this population, we will longitudinally track reproductive health of participants, including menstrual history, pregnancy rate, and biological (serum) markers of ovarian function. The FMR1 pre-mutation may also be associated with specific general health risks, such as hypertension, thyroid disease, neurological disorders, and psychiatric disorders. A patient registry will also allow us to track development of these and other common medical conditions to determine if women with the FMR1 pre-mutation have increased health risks. Currently, there are no screening guidelines regarding reproductive or general health for women who carry the FMR1 pre-mutation, and observations from longitudinal data will help to develop such guidelines. Finally, standardized guidelines for genetic counseling of women with the FMR1 pre-mutation regarding genetic risk to their children do not exist, and data collected in this study will enable this.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Women ages 18 and older
  2. FMR1 CGG repeats numbering between 55 and 199, as determined by standard Southern blot and PCR techniques.

EXCLUSION CRITERIA:

1. Males
2. Children
3. Women who do not have an FMR1 pre-mutation (CGG repeat number <55 or >199)
4. Inability to make personal medical decisions

CRITERIA FOR SCREENING FOR THE FMR1 PRE-MUTATION:

1. Family history of Fragile X syndrome or mental retardation
2. Personal or family history of primary ovarian insufficiency (or POF or premature menopause )
3. Personal or famiy history of tremor ataxia syndrome or Parkinson s disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-08-05; Study Completion 2013-05-31

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence M Nelson, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nelson LM. Clinical practice. Primary ovarian insufficiency. N Engl J Med. 2009 Feb 5;360(6):606-14. doi: 10.1056/NEJMcp0808697. PMID 19196677
- [Background] Hagerman RJ, Hagerman PJ. The fragile X premutation: into the phenotypic fold. Curr Opin Genet Dev. 2002 Jun;12(3):278-83. doi: 10.1016/s0959-437x(02)00299-x. PMID 12076670
- [Background] Wittenberger MD, Hagerman RJ, Sherman SL, McConkie-Rosell A, Welt CK, Rebar RW, Corrigan EC, Simpson JL, Nelson LM. The FMR1 premutation and reproduction. Fertil Steril. 2007 Mar;87(3):456-65. doi: 10.1016/j.fertnstert.2006.09.004. Epub 2006 Oct 30. PMID 17074338